CLINICAL TRIAL: NCT01102114
Title: A Second Phase 3, Multi-Center, Randomized, Double-Blind, Placebo-Controlled Study to Assess Efficacy, Immunogenicity and Safety of 3'-Aminomethylnicotine-P. Aeruginosa r-Exoprotein A Conjugate Vaccine (NicVAX) as an Aid to Smoking Cessation
Brief Title: A Second Study of NicVAX/Placebo as an Aid for Smoking Cessation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nabi Biopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Nabi-4515
Record Dates: First submitted 2010-03-17; First posted 2010-04-12 (Estimated); Last update posted 2012-05-09 (Estimated); Status verified 2012-05

CONDITIONS: Smoking Cessation
Keywords: Smoking Cessation; NicVAX; Smoking Vaccine; Smoking Abstinence; Smoking; Tobacco Cessation
MeSH Terms: conditions — Smoking Cessation; Smoking; Tobacco Use Cessation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo Vaccine (Placebo Comparator)
  Interventions: Biological: Placebo Vaccine
- NicVAX Vaccine (Experimental)
  Interventions: Biological: NicVAX Vaccine

INTERVENTIONS:
Biological: NicVAX Vaccine — NicVAX vaccine given 6 times over 6 months
  Arms: NicVAX Vaccine
Biological: Placebo Vaccine — Placebo vaccine given 6 times over 6 months
  Arms: Placebo Vaccine

SUMMARY:
The purpose of this study is to evaluate NicVAX as an aid to smoking cessation for long term abstinence.

ELIGIBILITY:
Inclusion Criteria:

* Current smoker who smokes at least 10 cigarettes a day during the past year and wants to quit smoking.
* Smokers who are in good general health.

Exclusion Criteria:

* Prior exposure to NicVAX or any other nicotine vaccine.
* Use of systemic steroids.
* Cancer or cancer treatment in the last 5 years.
* HIV infection.
* History of drug or alcohol abuse or dependence within 12 months.
* Significant cardiovascular, hepatic, renal, psychiatric and/or respiratory disease.
* Inability to fulfill all visits for approximately 52 weeks.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2010-03; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Evaluate NicVAX as an aid to smoking cessation for long term abstinence (by subject self-report and carbon monoxide confirmation). | One year

SECONDARY OUTCOMES:
Evaluate abstinence rates at multiple intervals (by subject self-report and carbon monoxide confirmation). | One year
Evaluate safety based on adverse events. | One year
Evaluate immunology based on serum antibody concentration. | One year
Evaluate withdrawal symptoms, smoking satisfaction, cigarette consumption and nicotine dependence (based on subject self-report). | One year

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Nabi Biopharmaceuticals
Locations (25):
- United States (25):
  - NicVAX Investigator, Encino, California
  - NicVAX Investigator, Los Alamitos, California
  - NicVAX Investigator, Denver, Colorado
  - NicVAX Investigator, New Haven, Connecticut
  - NicVAX Investigator, Brooksville, Florida
  - NicVAX Investigator, Orlando, Florida
  - NicVAX Investigator, Pembroke Pines, Florida
  - NicVAX Investigator, Tampa, Florida
  - NicVAX Investigator, Indianapolis, Indiana
  - NicVAX Investigator, Wichita, Kansas
  - NicVAX Investigator, Metairie, Louisiana
  - NicVAX Investigator, Annapolis, Maryland
  - NicVAX Investigator, Milford, Massachusetts
  - NicVAX Investigator, East Lansing, Michigan
  - NicVAX Investigator, Rochester, Minnesota
  - NicVAX Investigator, Jackson, Mississippi
  - NicVAX Investigator, Omaha, Nebraska
  - NicVAX Investigator, Buffalo, New York
  - NicVAX Investigator, Cincinnati, Ohio
  - NicVAX Investigator, Mt. Pleasant, South Carolina
  - NicVAX Investigator, Knoxville, Tennessee
  - NicVAX Investigator, Nashville, Tennessee
  - NicVAX Investigator, Houston, Texas
  - NicVAX Investigator, Salt Lake City, Utah
  - NicVAX Investigator, Charleston, West Virginia